CLINICAL TRIAL: NCT03937947
Title: Traumatic Brain Injury Associated Radiological Deep Venous Thrombosis Incidence and Significance
Brief Title: Traumatic Brain Injury Associated Radiological DVT Incidence and Significance Study
Acronym: TARDIS
Status: Completed | Type: Observational
Sponsor: NHS Lothian (Other Government)
Responsible Party: Principal Investigator, Jonathan Rhodes, Consultant in Intensive Care and Anaesthesia, NHS Lothian
Other Study IDs: AC18105; WKR0-2018-0020 (Other Grant/Funding Number: British Journal of Anaesthesia); WKR0-2018-0020 (Other Grant/Funding Number: Neuro Anaesthesia and Critical Care Society)
Record Dates: First submitted 2019-04-26; First posted 2019-05-06 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-09

CONDITIONS: Traumatic Brain Injury; Deep Vein Thrombosis; Acute Lung Injury; Ventilator Associated Pneumonia
MeSH Terms: conditions — Brain Injuries, Traumatic; Venous Thrombosis; Acute Lung Injury; Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Whilst deep vein thrombosis (DVT) is common following traumatic brain injury (TBI), optimal timing and safety of pharmacological prophylaxis is uncertain. Paradoxically the harm associated with the occurrence of is also unclear.

This study is an observational pilot that aims to define the incidence of proximal DVT in patients with moderate to severe TBI. It seeks prospectively to determine if there is an association between DVT and outcome. It also seeks to explore possible associations between the occurrence of DVT and the incidence of lung injury and/or ventilator associated pneumonia.

DETAILED DESCRIPTION:
Deep Venous Thrombosis (DVT) is common following trauma and patients with TBI are at increased risk. In studies of TBI that screened for DVT in the proximal lower limb veins, the incidence is between 14 and 18%. Pharmacological thromboprophylaxis (PT) may be effective in reducing the incidence of DVT following TBI. However, there is a reluctance to commence it due to concerns about the risk of intracranial haematoma expansion and contusion enlargement. PT is therefore often delayed, exposing patients to potential risks and complications of DVT. Recent systematic reviews could not answer the question of when to commence PT as no high quality randomised controlled trials addressing this question have been conducted. The latest edition of the Brain Trauma Foundation Guidelines could not make a recommendation on this issue . A Delphi exercise involving the investigator's network of United Kingdom(UK) Eurotherm3235 study centres found that the leading concern of specialists in UK neurocritical care, that they felt required further study, was when to commence PT following moderate to severe TBI.

Paradoxically however, despite these concerns over the use of PT in this population of patients, evidence of harm associated with the confirmed presence of proximal DVT is not yet convincing. This has additional significance as without clear evidence of harm associated with DVT complicating TBI, trials to address the questions of safety and efficacy of earlier use of PT are difficult to design and unlikely to attract the necessary funding.

From a search of a trauma registry of patients at risk of DVT who underwent venous screening, in TBI patients the occurrence of DVT was associated with increased ventilator days (Mean (SD), 18.0 (14.9) vs. 9.3 (7.9) days for DVT vs. no DVT, p=0.014) and ICU length of stay (23.0 (14.5) vs. 13.1 (9.8) days for DVT vs. no DVT, p=0.006). Similar results were seen in a post hoc analysis of the EPO TBI trial. This was a randomised controlled trial (RCT) of the effect of erythropoietin (EPO) verses placebo on outcome following TBI. Repeated lower limb screening for the presence of DVT was conducted as part of the protocol. Both ventilator days (Median (IQR) 11 (6-17) vs. 8 (4-14) days for DVT vs. no DVT, p<0.001) and ICU length of stay (17 (11-22) vs. 12 (6-19) days DVT vs. no DVT, p<0.001). Good neurological outcome at 6 months was significantly less frequent in those that developed DVT (45.4 vs. 57.9% DVT vs. no DVT, p=0.01). Whilst these findings are clinically important they are the result of retrospective and post hoc analysis. They therefore require to be prospectively validated if they are to be accepted.

One possible explanation for an increase in ventilator dependency and ICU length of stay could be the occurrence of undiagnosed pulmonary emboli causing acute lung injury (ALI). The occurrence of ventilation perfusion mismatching, deterioration in arterial partial pressure: fraction inspired oxygen ratio (PaO2:FiO2) and radiological changes on chest x-ray, being interpreted as evidence of pulmonary infection. This is supported by local audit data from June to October 2017 which found that 37% of brain injured patients had a clinical diagnosis of ventilator associated pneumonia (VAP) and were treated with antibiotics but lacked subsequent microbiological confirmation. It is also possible that small pulmonary emboli might predispose to pulmonary infection, explaining why the incidence of ventilator associated pneumonia (VAP) remains high in this population (40%, in the same local audit) despite the adoption of measures which have lowered VAP rates in other critically ill patient groups.

Lung Brain "cross-talk" could link evidence of ALI to a negative impact on neurological outcome in these patients. A disproportionate increase in mortality in patients with TBI and ALI has been reported. This was greatly in excess of deaths attributable to pulmonary dysfunction. Similarly, in animal models, ALI was found to be associated with cognitive impairment, and biomarker/histological evidence of neuronal injury.

This is a prospective, potentially multi centre, observational pilot study that aims to determine the incidence of DVT after TBI. Patients admitted to an ICU within 72 hours of suffering a TBI will be eligible for inclusion. The study will run for 2 years with a 16 month recruitment period. Based on current activity in Edinburgh the investigators estimate that 50 to 60 patients will be eligible for recruitment over the course of the study. In order to ensure satisfactory recruitment, the investigators will also approach centres that have expressed an interest.

Once consent is obtained for the patient to be enrolled in the study, a compression ultrasound scan (USS) of both legs will be carried out as soon as possible so that the first USS is completed within 72 hours of injury. USS will be repeated on alternate days up to Day 10 from injury. Daily data collection will include information on the use of mechanical and pharmacological thromboprophylaxis, ventilator dynamics including FiO2 and PaO2, chest X ray reports, clinical and microbiological diagnosis of ventilator associated pneumonia, ventilator days and ICU and hospital length of stay. The Modified Oxford Handicap Scale will be completed for all patients on day 28, hospital discharge or death whichever is sooner Patients will then be followed up at 6 months by the study team, at which time an extended Glasgow Outcome Scale Questionnaire will be completed.

An amendment to the protocol is also being prepared to include assessment of blood coagulation by standard laboratory testing and viscoelastic methods.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 16 years
2. Admission to critical care
3. moderate/severe, non-penetrating traumatic brain injury
4. Abnormal brain CT Scan
5. Post resuscitation Glasgow coma score (GCS) ≤12, or GCS motor component ≤5
6. Able to complete consent and first USS within 72 hours of injury

Exclusion Criteria:

1. Normal brain CT scan
2. Unlikely to survive for the next 24 hours in the opinion of the ICU Consultant or Consultant Neurosurgeon treating the patient
3. Contra indication to normal prophylactic measures, including heparin, were indicated
4. Known blood clotting disorder or thrombophilia
5. Significant pelvic or lower limb trauma
6. Malignancy
7. Pregnancy or recently post-partum

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults with moderate to severe TBI requiring critical care support.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-09-28 (Actual); Primary Completion 2023-09-24 (Actual); Study Completion 2023-09-24 (Actual)

PRIMARY OUTCOMES:
Incidence of proximal DVT by compression ultra sound | within 72 hours of injury until day 10 post injury.
  Alternate day compression ultra sound

SECONDARY OUTCOMES:
Incidence of Acute Lung Injury | Up to 10 days post injury
  PaO2:FiO2 <300 mmHg
Incidence of Ventilator Associated Pneumonia | Up to 10 days post injury
  Hospitals in Europe Link for Infection Control through Surveillance/European Centre for Disease Control and Prevention (HELICS/ESDC) criteria
Ventilator days in ICU | From day of injury until death whilst receiving ventilatory support or no longer requiring actively ventilation or respiratory support greater than the provision of continuous positive airways pressure (CPAP) via a tracheostomy, upto 6 months.
  Days or part off that respiratory support was provided via endotracheal tube or tracheostomy
Length of Stay in ICU | From day of injury until day of death or discharge from ICU to a step down unit providing level 1 care or lower, upto 6 months.
  Days or part off in ICU
Hospital Length of Stay | From day of injury until day of death or hospital discharge to a rehabilitation facility, nursing facility, or patient's home, assessed upto 6 months.
  Days or part of in hospital
Modified Oxford Handicap Score | To be completed on day 28 after injury, hospital discharge or death whichever occurs first.
  Functional Outcome- a score of 0 indicates no symptoms, 1 minor symptoms, 2 some restriction, 3 dependent, 4 fully dependent, and 5 death.
Extended Glasgow Outcome Scale | 6 months
  Functional Outcome - a score of 1 indicates death, 2 vegetative state, 3 lower severe disability, 4 upper severe disability, 5 lower moderate disability, 6 upper moderate disability, 7 lower good recovery , 8 upper good recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- Intensive Care Unit, Western General Hospital, Edinburgh, Midlothian, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data at present.